CLINICAL TRIAL: NCT06629428
Title: Effects of Ublituximab on Unperturbed and Perturbed Ambulatory Functions in People With Relapsing Multiple Sclerosis
Brief Title: Effects of Ublituximab on Motor Functions in Multiple Sclerosis
Acronym: U-PACE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Atlanta Neuroscience Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H25013
Record Dates: First submitted 2024-09-19; First posted 2024-10-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: ublituximab; gait function; disease progression; perturbed walking; Cognition
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Disease Progression | interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ublituximab (Experimental): This arm will receive a 48-week ublituximab treatment.
  Interventions: Drug: Ublituximab

INTERVENTIONS:
Drug: Ublituximab — The participants will receive 48 weeks of treatment with ublituximab.

SUMMARY:
The purpose of this study is to test if ublituximab changes walking functions and fall risk in people with relapsing multiple sclerosis (RMS). Twenty-five qualified people with RMS will undergo a 48-week ublituximab treatment. Before, 24 weeks into, and after the treatment, their ambulatory function, disability status, and cognition will be assessed. Additionally, they will experience large-scale slip perturbations on a treadmill under the protection of a safety harness at the last assessment. The outcome measures will be compared across the assessments to examine the effects of ublituximab on improving their walking function, disability status, cognition, and the responses to the unexpected slip perturbation.

DETAILED DESCRIPTION:
The primary objective of this single-arm and pretest-posttest study will be to examine the effects of treatment with ublituximab on ambulatory functions during unperturbed walking and large-scale gait slips (dynamic gait stability and slip-fall) among people with relapsing MS over a 12-month treatment period. Additionally, the effects of ublituximab on disease progression and cognitive functions will be evaluated.

Twenty-five qualified people with relapsing multiple sclerosis (RMS) will be enrolled to this study. Before the treatment, their ambulatory functions during regular walking will be assessed in terms of their spatiotemporal gait parameters. This assessment is considered the baseline test. Their disease progression will be evaluated by the neurological exam and serum neurofilament light chain. Their cognitive function will be tested by the Montreal Cognitive Assessment. Then, they will undergo the 48-week ublituximab treatment. At the mid-point of the treatment period, they will attend another assessment session, which is identical to the baseline session. Immediately after the 48-week treatment, the same assessments will be executed again as the baseline test. In addition, all participants will experience repeated unexpected slip perturbations while walking on a treadmill under the protection of a full-body safety harness. Their response to the the slips will be quantified by their dynamic balance, reaction times of the lower leg muscles, and adaptation rate to the repeated slips.

All the measurements will be analyzed to identify the effects of ublituximab on ambulatory functions, disease progression, and cognitive status of people with relapsing multiple sclerosis.

Our findings will potentially lead to earlier adoption of this highly efficacious disease-modifying treatment and thus likely improve long-term patient care outcomes. This study will uncover how ublituximab impacts ambulatory function and mobility among people with relapsing MS. This will augment our current understanding of ublituximab which focuses on the aspect of the disease progression. Given mobility is critical for people with MS to maintain their employment, independence, participation in social events, and thus the quality of life, this study will have great potential to scientifically enhance our scientific understanding of effects of ublituximab and to clinically improve patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, informed consent and to be compliant with the schedule of protocol assessments.
2. Ages between 18 and 55 years old at screening.
3. Clinically confirmed active, relapsing forms of MS based on the revised McDonald criteria.
4. Can walk at least 25 feet independently with or without assistive devices at screening.
5. Can stand independently for at least 30 seconds.
6. Not pregnant at screening and throughout the study.

   * A negative urine or serum pregnancy test must be available for premenopausal women and for women < 12 months after the onset of menopause at screening, unless they have undergone surgical sterilization.
   * Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use one method of contraception with a failure rate of < 1% per year or a barrier method supplemented with spermicide. Contraception must continue for the duration of study treatment and for at least 6 months after the last dose of study treatment.

     * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of the ovaries and/or uterus).
     * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tube ligation, male sterilization, established hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
     * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception.
     * Examples of barrier methods supplemented with the use of spermicide include male or female condom, vaginal ring, cap, diaphragm, or sponge.
7. No other neurological conditions and recent musculoskeletal injuries.
8. Can read and understand English.
9. No significant cognitive impairment.

Exclusion Criteria:

Basic Exclusion Criteria

1. History of MS types other than relapsing MS at screening (such as primary-progressive MS, inactive SPMS).
2. History of life-threatening infusion reaction on ublituximab, any of its ingredients, or prior anti-clusters of differentiation 20 (CD20) therapy.
3. Hypersensitive to any of the ingredients of ublituximab.
4. Do not understand English.

   Exclusions Related to General Health
5. Pregnancy or lactation.
6. Have any other known neurological diseases which may mimic MS, including but not limited to: Neuromyelitis optica, Lyme disease, untreated vitamin B12 deficiency, neurosarcoidosis, and cerebrovascular disorders.
7. History of clinically significant central nervous system (CNS) trauma (e.g., traumatic brain injury, cerebral contusion, spinal cord compression, etc.).
8. History of liver disease.
9. Active hepatitis B virus (HBV) confirmed by positive results for Hepatitis B surface antigen (HBsAg) and anti-HBV tests.
10. Current evidence or known history of clinically significant infection.
11. Suffering from coexisting psychiatric disorders, neurological disorders, or severe medical illness.
12. Current severe depression and/or suicidal ideation.
13. Significant cognitive impairment (Montreal Cognitive Assessment or Montreal Cognitive Assessment (MoCA) score < 24).
14. New onset, unstable orthopedic comorbid diagnoses (within 3 months and uncontrolled).
15. History or currently active primary or secondary immunodeficiency.
16. Receipt of a live vaccine within 6 weeks before baseline.
17. Skin is allergic to transparent double-side tapes.
18. Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
19. History or currently active primary or secondary immunodeficiency.
20. Lack of peripheral venous access.
21. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
22. Significant or uncontrolled somatic disease or any other significant disease that may preclude a patient from participating in the study.
23. Congestive heart failure (NYHA III or IV functional severity).
24. Known active bacterial, viral, fungal, mycobacterial infection or other infection, excluding fungal infection of nail beds.
25. Infection requiring hospitalization or treatment with i.v. antibiotics within four weeks prior to baseline visit or oral antibiotics within two weeks prior to baseline visit.
26. History or known presence of recurrent or chronic infection (e.g., hepatitis B or C, HIV, syphilis, tuberculosis).
27. History of progressive multifocal leukoencephalopathy (PML).
28. History of malignancy, including solid tumors and hematological malignancies, except basal cell carcinoma, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix of the uterus that has been previously completely excised with documented clear margins.
29. History of alcohol or drug abuse within 24 weeks prior to baseline.
30. History or laboratory evidence of coagulation disorders.

    Exclusions Related to Medications
31. Receipt of any live of live-attenuated vaccines within 4 weeks prior to first drug product administration.
32. Treatment with any investigational agent within 24 weeks of screening (Visit 1) or five half-lives of the investigational drug (whichever is longer).
33. Systemic corticosteroid therapy within 4 weeks prior to screening.
34. Any previous treatment with alemtuzumab (Campath), anti-cluster of differentiation 4 (CD4), cladribine, mitoxantrone, daclizumab, tecfidera (BG12), teriflunomide, laquinimod, total body irradiation or bone marrow transplantation.
35. Treatment with cyclophosphamide, azathioprine, mycophenolate mofetil (MMF), cyclosporine, methotrexate, or natalizumab within 24 months prior to screening.
36. Treatment with intravenous immunoglobulin within 12 weeks prior to baseline.
37. Treatment with anti-CD20 or other B cell-directed treatment.

    Exclusions Related to Motor Function
38. Cannot walk at least 25 feet and stand for at least 30 seconds independently.
39. Weak or blind vision may impair their ability to walk.

    Exclusions Related to Musculoskeletal, Cardiovascular, and Orthopedic Conditions
40. Broken bones as an adult in the past year.
41. Have received neurological treatment, such as Botox, in the past six months.
42. Heart attack, angioplasty, or coronary artery bypass graft in the past six months.
43. Congestive heart failure (NYHA III or IV functional severity).
44. Surgery on back, hip, shoulder, or total joint replacement of hip or knee joint less than two years ago.
45. Respiratory conditions (lung cancer, bronchitis, emphysema, asthma, shortness of breath) not under regular medical care or the patient is medically unstable.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
slip-fall | 48 weeks
  The outcome of a slip trial will be deemed a fall if the peak load cell force exceeds 30% of the body weight.
Dynamic gait stability during slip | 48 weeks
  For a slip, dynamic gait stability will be calculated at two events: the slipping foot touchdown and the recovery foot liftoff.

SECONDARY OUTCOMES:
Dynamic gait stability during walking | weeks 0, 24, and 48
  Dynamic gait stability during walking will be calculated based on the theoretical framework of Feasible Stability Region.
Spatiotemporal gait parameters during walking | Weeks 0, 24, and 48
  The following parameters will be determined: gait speed, step length, step width, step time, and cadence. These measurements will be used to quantify our participants' ambulatory functions.
Leg muscle strength | Weeks 0, 24, and 48
  The maximum voluntary muscle strength will be assessed during maximum voluntary contractions at bilateral knee and ankle joints on an isokinetic dynamometer.
Leg Muscle Activities | Weeks 0, 24, and 48
  The surface electromyography activity from four muscles on each leg: the tibialis anterior (TA), medial gastrocnemius (MGAS), vastus lateralis (VLAT), and biceps femoris long head (BFLH), will be recorded.
Sway index | Weeks 0, 24, and 48
  It is measured when a patient is standing still for 30 seconds under four conditions: eyes open on a firm surface, eyes closed on a firm surface, eyes open on a foam pad, and eyes closed on a foam pad.
Stability index | Weeks 0, 24, and 48
  The overall stability index during stance will be determined based on the center of pressure trace calculated from the ground reaction forces.
Expanded Disability Status Scale | Weeks 0, 24, and 48
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability.
Multiple Sclerosis Functional Composite | Weeks 0, 24, and 48
  The three dimensions of the multiple sclerosis functional composite (MSFC) score: lower extremity motor function, upper extremity motor function, and cognitive function, will be collected based on the guidelines and forms provided by the National MS Society.
Prospective falls | Through study completion, an average of 1 year
  Participants in both groups will keep track of any falls they experience in the 12 months after the baseline evaluation using the falls questionnaire.
Serum neurofilament light chain | Weeks 0, 24, and 48
  The serum neurofilament light chain level serves as a biological marker of neuronal damage and disease progression. It will be collected for all participants in this project.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - Atlanta Neuroscience Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhle J, Plavina T, Barro C, Disanto G, Sangurdekar D, Singh CM, de Moor C, Engle B, Kieseier BC, Fisher E, Kappos L, Rudick RA, Goyal J. Neurofilament light levels are associated with long-term outcomes in multiple sclerosis. Mult Scler. 2020 Nov;26(13):1691-1699. doi: 10.1177/1352458519885613. Epub 2019 Nov 4. PMID 31680621
- [Background] Yang F, Bhatt T, Pai YC. Generalization of treadmill-slip training to prevent a fall following a sudden (novel) slip in over-ground walking. J Biomech. 2013 Jan 4;46(1):63-9. doi: 10.1016/j.jbiomech.2012.10.002. Epub 2012 Nov 8. PMID 23141636
- [Background] Yang F, Pai YC. Automatic recognition of falls in gait-slip training: Harness load cell based criteria. J Biomech. 2011 Aug 11;44(12):2243-9. doi: 10.1016/j.jbiomech.2011.05.039. Epub 2011 Jun 21. PMID 21696744
- [Background] Carpenter MR, Carpenter RL, Peel J, Zukley LM, Angelopoulou KM, Fischer I, Angelopoulos TJ, Rippe JM. The reliability of isokinetic and isometric leg strength measures among individuals with symptoms of mild osteoarthritis. J Sports Med Phys Fitness. 2006 Dec;46(4):585-9. PMID 17119524
- [Background] Simoneau GG. Kinesiology of walking. In: Neumann D. A., editor. Kinesiology of the Musculoskeletal System: Foundations of Physical Rehabilitation. St. Louis: Mosby; 2010. p. 636.